CLINICAL TRIAL: NCT02452905
Title: A Phase II Double-blind Randomised, Placebo-controlled Clinical Trial of Oral Nitazoxanide for the Treatment of Bronchiolitis in Infants Presenting to Hospital Emergency Departments
Brief Title: Finding Better Treatment of Bronchiolitis: A Clinical Trial of Oral Nitazoxanide for the Treatment of Bronchiolitis in Infants Presenting to Hospital Emergency Departments
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The drug manufacture were unable to produce liquid formulation of the IMP within a reasonable time frame so the funding was relinquished.
Sponsor: Telethon Kids Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVID/2014-02
Record Dates: First submitted 2015-05-12; First posted 2015-05-25 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitazoxanide (Active Comparator): Nitazoxanide 7.5mg/kg oral/nasogastric/nasoenteric tube three times per day for five days.
  Interventions: Drug: Nitazoxanide
- Placebo (Placebo Comparator): The placebo is identical to the active drug described above except that it does not contain the active compound nitazoxanide. It is reconstitutes, administered and dosed as per the active study drug.
  Interventions: Drug: Placebo (for Nitazoxanide)

INTERVENTIONS:
Drug: Nitazoxanide
  Other Names: Alinia
  Arms: Nitazoxanide
Drug: Placebo (for Nitazoxanide)
  Arms: Placebo

SUMMARY:
Bronchiolitis is an extremely common cause of respiratory illness in infants caused by viral infection.This study evaluates whether treatment with nitazoxanide (NTZ) reduces the duration and severity of respiratory symptoms caused by bronchiolitis. Half of the participants will receive NTZ while the other half will receive a placebo.

DETAILED DESCRIPTION:
Nitazoxanide (NTZ) is a novel anti-infective medication that is licenced for use in the United States (US), including in children and infants for treating some infections. It is in the thiazolide class of antimicrobials and has been shown to have in vitro and/or clinical activity against a broad spectrum of pathogens, including a range of viruses, parasites and bacteria.

This study will determine whether NTZ is an effective empirical treatment for bronchiolitis. It will also help us to understand what effect NTZ has on the amount of virus present and how viral load changes over the course of the disease. If this study shows that NTZ is a useful treatment, then a larger study will be conducted enrolling infants that present to primary care facilities.

ELIGIBILITY:
Inclusion Criteria:

* Aged greater than or equal to 1 month to less than or equal to 12 months
* Diagnosed with bronchiolitis by the assessing doctor
* Parent/legally responsible carer has provided informed consent for their infant/child to participate in the study
* Parent/legally responsible carer able and willing to comply with the requirements of the protocol
* Parent/legally responsible carer willing to attend a study follow up visit on study day 3 if their infant/child has previously been discharged from hospital
* Parent/legally responsible carer willing to allow other parties involved in the treatment of his or her child (including the general practitioner, paediatrician, hospital medical and nursing staff, community clinic staff) to be notified of participation in the trial
* Infants and children whose parent is willing to allow the study team to obtain an interim medical history from the participants electronic medical records (including immunisation records) and/or from the participants general practitioner or other medical professional for the period from enrolment to study day 180

Exclusion Criteria:

* Presence of symptoms of bronchiolitis (breathing difficulty, difficulty feeding, cough, poor feeding) for greater than or equal to 48 hours at the time of enrolment
* Born at gestational age of less than 32 weeks
* Has a history of any condition associated with risk of severe bronchiolitis including (significant cardiovascular disease, including congenital heart disease, significant respiratory disease including chronic lung disease, Trisomy 21, significant neurological disease including history of seizure disorder, significant impairment/alteration of the immune system including congenital immunodeficiency or any other disorder considered relevant by a medically qualified investigator
* Requiring admission to intensive care unit at enrolment
* Clinical suspicion of illness other than bronchiolitis
* Contraindication to the study drug or placebo (hypersensitivity), medical treatment with medication which in the opinion of the admitting team would make the child unsuitable for the study
* Receipt of investigational drug/vaccine, other than the drugs used in the study within 30 days prior to receiving the first dose of NTZ or their planned use during the study period until 1 month after the administration of the final dose of NTZ
* Previously enrolled in the study
* Parent less than 18 years of age

TEMPORARY EXCLUSION CRITERIA

* Receipt of an anti-viral medication within the previous 7 days
* Inability to tolerate either the oral or nasogastric route (e.g. ileus)
* Any systemic corticosteroid (or equivalent) treatment in 14 days prior to enrolment

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2017-10 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Severity of respiratory distress | Up to day 4
  The calculation of a Respiratory Assessment Change Score (RACS) by the use of the Respiratory Distress Assessment Instrument (RDAI) from baseline (day 1) to study day 4 adjusted for the standardised change in respiratory rate with points being assigned by change increments of 10% Internal reliability and responsiveness of the RACS as a measure of respiratory distress in infants has been previously demonstrated and it correlates well with other measures of respiratory distress

SECONDARY OUTCOMES:
Nasopharyngeal excretion of Respiratory Syncytial Virus (RSV) | Up to 72 hours
  The change in nasopharyngeal viral excretion as measured by Polymerase Chain Reaction (PCR)
Duration of parent reported solicited symptoms associated with bronchiolitis during and after treatment | Up to day 7
  The time until the severity of ALL solicited symptoms associated with bronchiolitis (loss of appetite, activity level, respiratory effort and irritability) have first been assessed as mild or normal from the day of randomisation to the end of study day 7
Actual duration of hospital admission for any reason | Participants will be followed for the duration of hospital stay, an expected average of 1 to 3 days.
  The period of time for which hospitalisation is required for any medical reason
Need for interventional supportive medical care | Up to day 7
  The use of oxygen therapy, supportive ventilation, admission to the Intensive Care Unit (ICU) and supportive hydration therapy (NG or IV). Duration of use is calculated from the calendar day of randomisation to the date of cessation
Severity of parent reported solicited symptoms associated with bronchiolitis during and after treatment | Up to day 7
  The time until the severity of ALL solicited symptoms associated with bronchiolitis (loss of appetite, activity level, respiratory effort and irritability) have first been assessed as mild or normal from the day of randomisation to the end of study day 7
Duration of interventional supportive medical care | Up to day 7
  The use of oxygen therapy, supportive ventilation, admission to the Intensive Care Unit (ICU) and supportive hydration therapy (NG or IV). Duration of use is calculated from the calendar day of randomisation to the date of cessation

OTHER OUTCOMES:
Occurrence of adverse events attributed to the study treatment | Participants will be followed for the duration of enrolment and up to 180 days post completion
  The occurrence of adverse events attributed to the study treatment
Recurrent bronchiolitis requiring health care assessment and /or intervention | Within 6 months of enrolment
  Recurrent bronchiolitis requiring health care assessment and/or intervention
Prolongation of bronchiolitis | Up to 180 days post completion
  Prolongation of bronchiolitis beyond day 7 after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Claire WADDINGTON, BMBS MSc MRCP (UK) DPhil, Principal Investigator — Telethon Kids Institute
Locations (1):
- Telethon Kids Institute, Perth, Western Australia, Australia